CLINICAL TRIAL: NCT02380209
Title: An Early Phase Clinical Trial to Evaluate the Feasibility of CEST MRI in Patients With Early Stage Breast Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI has terminated study as the sequencing on patients and volunteers didn't yield the results expected. PI has no plans for scholarly/scientific presentations.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1406349968
Record Dates: First submitted 2015-01-09; First posted 2015-03-05 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; CEST MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — iopromide; Iopamidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Optimization (Experimental): CEST MRI of the breast for estimation of tumor pH.
  Interventions: Other: CEST MRI

INTERVENTIONS:
Other: CEST MRI — CEST MRI will be performed on patients prior to surgical resection of their tumor
  Other Names: iopromide; Ultravist; Isovue

SUMMARY:
Evaluate the feasibility of translating preclinical Chemical Exchange Saturation Transfer (CEST) MRI protocol designed to estimate tumor extracellular pH (pHe) to a clinical MRI scanner in women with early stage breast cancer. Assays are used to quantify tumor acidosis.

DETAILED DESCRIPTION:
Those involved in the treatment of patients with breast cancer have pioneered the field of personalized cancer therapy through the use of targeted therapies and their associated biomarkers. Assays to quantify tumor acidosis and hypoxia are hypothesized to potentially represent such biomarkers. However there is currently no gold standard for measuring either.

This trial will evaluate the feasibility of translating preclinical Chemical Exchange Saturation Transfer (CEST) MRI protocol designed to estimate tumor extracellular pH (pHe), to a clinical MRI scanner in women with early stage breast cancer. This trial will generate preliminary data regarding the feasibility of this imaging technique. If successful, in future studies CEST MRI may serve as an imaging biomarker for acidosis and hypoxia.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed infiltrating ductal carcinoma (IDC) of the breast
* >= 1.0 cm primary tumor
* Calculated creatinine clearance >= 50 mL/min
* Willing and able to provide informed consent
* Age ≥ 18 years
* ECOG performance status 0-2
* Informed of the investigational nature of this study

Exclusion Criteria:

* Allergy to iodinated contrast agent
* Use of metformin, aminoglycosides, other nephrotoxic medications, or daily use of NSAIDs
* Diabetes mellitus
* History of severe claustrophobia
* Presence of electrically, magnetically, or mechanically activated implants including cardiac pacemakers, cochlear implants, magnetic surgical clips or prosthesis that would preclude MRI
* Use of > 1 antihypertensive drug
* Pregnancy or breastfeeding
* Paraproteinemia syndromes or multiple myeloma
* Collagen vascular disease
* Active hyperthyroidism
* Active pharmaceutical treatments for cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
pH measurement of the tumor will be measured by the CEST MRI. | 2 weeks
  pH estimate of the tumor

SECONDARY OUTCOMES:
Correlate tumor pH as estimated by CEST MRI with protein and RNA based markers for acidosis and hypoxia. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at UMC North, Tucson, Arizona, United States